CLINICAL TRIAL: NCT07195539
Title: CO2 Fractional Laser With Tranexamic Acid As An Effective Tool For Post Burn Hyperpigmentation.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Shumaila Dogar, Senior Registrar, King Edward Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 388/RC/KEMU
Record Dates: First submitted 2025-09-09; First posted 2025-09-26 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-06

CONDITIONS: Post Burn Hyperpigmentation
Keywords: fractional ablative laser; tranexamic acid; post burn hyperpigmentation
MeSH Terms: interventions — Lasers, Gas

STUDY DESIGN:
Intervention Model Description: same patient will be receiving both treatments on different parts.each participant act as their own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hyperpigmented lesion divided into halves and one for tranexamic acid one for saline (Experimental): this will be a split face study, each lesion will be divided into 2 halves one half will receive tranexamic acid spray while other will receive saline spray. each patient will act as his own control.
  Interventions: Other: Tranexamic Acid sprinkle with CO2 LASER

INTERVENTIONS:
Other: Tranexamic Acid sprinkle with CO2 LASER — tranexamin acid will be sprayed after CO2 LASER

SUMMARY:
It will be a case within control trial. After IRB approval patients presenting with more than 6 months old hyperpigmented burn scars will be included in this study.

All data (including age, gender, mode of burn) will be recorded on a proforma and standardized pre-intervention photographs will be taken. The hyperpigmented scar will be divided into two equal halves.One half will receive fractional CO2 wit TXA solution other half will receive fractional CO2 Laser with N/S solution.Thus allocation will be done randomly with the lottery method.

Total 3 sessions of LADD will be done with 1 month interval between each session. The following settings will be used: probe frequency 75Hz; Power range 12-15W; dwell time 300 micros-500 micros, stach 1-2 and spacing 900-1200m. The TXN solution will be prepared by mixing 250mg of TXA in 5ml of N/S creating a 5% TXN solution. Standardized photographs will again be taken 3 months after the 3rd session. The pre- and post-treatment photographs will be assessed by Skin Hyperpigmentation Index (SHI) using a smartphone dermatoscope adapter and an online calculator, freely available at: https://shi.skini magea nalys is.com, can be used. 15. Any complications during treatment will be noted and documented. Patient satisfaction wil be measured on a Likert scale of 1-5.

DETAILED DESCRIPTION:
TITLE:

CO2 FRACTIONAL LASER WITH TRANEXAMIC ACID AS AN EFFECTIVE TOOL FOR POST BURN HYPERPIGMENTATION.

INTRODUCTION Hyperpigmentation is one of the most common sequelae of burns and is due to dysregulation of normal wound healing after burn injury to skin1,2. The proinflammatory cytokine response after a burn stimulates melanocyte proliferation causing increased melanogenesis3. Patients with darker skin are more likely to have hyperpigmented scars. These cosmetically unappealing scars are even more concerning when they involve visible areas of the body, such as the face and hands.

Nonsurgical interventions to prevent or reduce hyperpigmentation of burn scars includes UV protection, hydroquinone application, silicone gel/sheet, nanofat grafting, cryotherapy, and laser and light therapy4. It has also been demonstrated that the earlier the intervention, the better the outcomes are likely to be.

Laser therapy has emerged as a minimally invasive intervention with short post-operative recovery5. Lasers are broadly categorized as ablative or non-ablative, and fractional or non-fractional. Ablative lasers such as the carbon-dioxide (CO2) and Erbium: Yag lasers are generally more effective, but pose a risk of adverse events such as infection, scarring and worsening of pigmentation6. Fractional photo-thermolysis, first described in 2004, leaves columns of non-treated areas between treated columns, thus allowing better wound healing7. Therefore, fractional lasers balance the efficacy of ablative lasers and the safety of non-ablative lasers. Fractional CO2 laser serves to increase dermal pliability, improve abnormal texture, reduce thickness and rehabilitate mature old scars8. A meta-analysis by Zhang et al demonstrated that fractional CO2 laser improved the appearance and pigmentation of post burn scars9.

Tranexamic acid (TXA) is a synthetic amino-acid derivative with hemostatic and anti-inflammatory properties. It works to decrease pigmentation through two mechanisms. Firstly, it reduces inflammatory melanogenesis by inhibiting the conversion of plasminogen to plasmin. Secondly, its causes activation of phagocytosis, leading to degradation of melanogenic enzymes10,11. It is in widespread use in the treatment of hyperpigmentation of melasma12.

Furthermore, laser-assisted drug delivery (LADD) techniques are gaining popularity. Fractional lasers create micro-columns that allows the drug to penetrate into the deeper dermis, and enhances the absorption of topically applied medication13.

The synergistic action of these individual treatments will have favorable outcomes in improving hyperpigmentation in burn scars14. Though there exists data to support this, there is a paucity of literature that specifically studies this effect in the South Asian population with Fitzpatrick skin types 3 and 4 OBJECTIVE; To compare the effects Laser assisted drug delivery of tranexamic acid, versus CO2 laser alone, in treating post burn hyperpigmentation in South Asian skin (Fitzpatrick type 3&4)

OPERATIONAL DEFINITION; POST BURN HYPERPIGMENTATION; Hyperpigmentation of skin after burn injury, it is more severe in dark-skinned individuals (Fitzpatrick III-VI) ABLATIVE LASER; Any laser that removes skin cells is known as ablative laser. FRACTIONAL LASER; It is a type of laser that targets a portion of skin at a time, leaving normal columns of skin

HYPOTHESIS: Fractional CO2 Laser assisted drug delivery of tranexamic acid will improve post burn hyperpigmentation to a greater degree than Laser alone in South Asian skin (Fitzpatrick III-IV).

SAMPLE SIZE:

Total of 30 patients will be enrolled. A p-value < 0.05 will be considered statistically significant.

Based on previous findings using the Skin Hyperpigmentation Index (SHI) in melasma patients (Heidemeyer et al., 2023), the estimated standard deviation of SHI scores is approximately 0.52. Assuming a mean difference of 0.5 units between treatment sides in a split-face design, and using a two-tailed paired t-test with 90% power and α = 0.05, a minimum of 19 participants is required to detect a statistically significant difference.

MATERIAL AND METHODS:

It will be a case within control trial. After IRB approval patients presenting with more than 6 months old hyperpigmented burn scars will be included in this study.

All data (including age, gender, mode of burn) will be recorded on a proforma and standardized pre-intervention photographs will be taken. The hyperpigmented scar will be divided into two equal halves.One half will receive fractional CO2 wit TXA solution other half will receive fractional CO2 Laser with N/S solution.Thus allocation will be done randomly with the lottery method.

Total 3 sessions of LADD will be done with 1 month interval between each session. The following settings will be used: probe frequency 75Hz; Power range 12-15W; dwell time 300 micros-500 micros, stach 1-2 and spacing 900-1200m. The TXN solution will be prepared by mixing 250mg of TXA in 5ml of N/S creating a 5% TXN solution. Standardized photographs will again be taken 3 months after the 3rd session. The pre- and post-treatment photographs will be assessed by Skin Hyperpigmentation Index (SHI) using a smartphone dermatoscope adapter and an online calculator, freely available at: https://shi.skini magea nalys is.com, can be used. 15. Any complications during treatment will be noted and documented. Patient satisfaction wil be measured on a Likert scale of 1-5.

Inclusion Criteria:

* Managed conservatively and healed within 3-4 weeks
* Age more than 18y
* Hyperpigmented Burn scar presenting after 6 months
* Patients with burn scar on face, neck, hands

Exclusion Criteria:

* Pregnant and breast feeding women
* Previous laser treatment
* Coagulation or platelet disorder
* Patients on anticoagulant medications/birth control pills
* DM/Connective tissue disorder
* Active viral infection
* History of malignancy/chemotherapy.

Data Analysis All data will be entered and analyzed using IBM SPSS (IBM Corp., Armonk, N.Y.) version 22.0. quantitative variables such as age will be given as mean. The qualitative variables such as gender, scar improvement and patient satisfaction will be calculated as frequency or percentage. Two tailed pair-t test will be used to compare the scar improvement between the two groups as well as compare scar improvement beween the genders and different age groups.

ELIGIBILITY:
Inclusion Criteria:• Managed conservatively and healed within 3-4 weeks

* Age more than 18y
* Hyperpigmented Burn scar presenting after 6 months
* Patients with burn scar on face, neck, hands

Exclusion Criteria:• Pregnant and breast feeding women

* Previous laser treatment
* Coagulation or platelet disorder
* Patients on anticoagulant medications/birth control pills
* DM/Connective tissue disorder
* Active viral infection
* History of malignancy/chemotherapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
improvement in hyperpigmentation | 3 months after completion of sessions
hyperpigmentation | 3months after completion of sessions
  Skin Hyperpigmentation Index will be used to determine improvement in hyperpigmentation.

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
we may not share it to conceal privacy of participants.

REFERENCES:
- [Background] Schaffrick L, Ding J, Kwan P, Tredget E. The dynamic changes of monocytes and cytokines during wound healing post-burn injury. Cytokine. 2023 Aug;168:156231. doi: 10.1016/j.cyto.2023.156231. Epub 2023 May 27. PMID 37247448
- See also: SHI will be used to measure improvement in hyperpigmentation — https://shi.skinimageanalysis.com/